CLINICAL TRIAL: NCT07119086
Title: Factors Associated With Hospitalization and Severity of Arbovirosis in the Indian Ocean
Acronym: ARB-OI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025/CHU/03; ID-RCB (Other Grant/Funding Number: 2025-A00359-40)
Record Dates: First submitted 2025-05-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Arbovirus Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patient with (Other): Blood samples and questionnaires
  Interventions: Biological: Biological samples; Other: Questionnaires

INTERVENTIONS:
Biological: Biological samples — Blood and urine samples
Other: Questionnaires — Quality of life questionnaires

SUMMARY:
Arboviroses, such as dengue, chikungunya and the Zika virus, represent a growing threat to public health in the Indian Ocean, but also in Europe and the rest of the world. Réunion has experienced several major epidemics, notably chikungunya in 2005-2006 and dengue since 2018, with a current resurgence of chikungunya. Mayotte was hit by a dengue epidemic in 2019, followed by a few cases of Rift Valley fever. The development of Zika could also affect this region.

Arboviruses, transmitted by hematophagous arthropods, require the coexistence of a reservoir and a vector. Dengue fever, transmitted by Aedes mosquitoes, is caused by four serotypes of dengue virus (DENV) from the orthoflavivirus family. Primary infection with one serotype confers lasting specific immunity, but only transient protection against the other serotypes. Chikungunya, caused by an alphavirus, now causes epidemics in major tropical areas. It is also transmitted by Aedes mosquitoes.

Arboviruses present four main clinical forms: algoeruptive, hemorrhagic, neurological and arthritic. Dengue fever is 75% asymptomatic, but can progress to a severe form, dengue hemorrhagic fever, characterized by increased vascular permeability and potentially fatal complications. Chikungunya causes a sudden onset of fever, polyarthralgia and maculopapular rash, with possible complications in newborns, the elderly and pregnant women.

Understanding the factors associated with hospitalization and the severity of these infections is crucial to improving patient management and optimizing medical resources. This cohort study aims to identify the clinical, demographic and environmental determinants influencing the severity of arbovirosis. By analyzing data from patients who have used a healthcare facility, we hope to establish risk profiles and severity criteria that may or may not be specific to each infection. The results will enable us to better understand the pathophysiology of these viruses, develop targeted prevention strategies and improve treatment protocols, thereby helping to reduce the morbidity and mortality associated with arboviroses in this region.

Due to the current chikungunya epidemic in La Réunion, this study will focus on the inclusion of patients affected by this arbovirosis as early as 2025. Its openness over the coming years will allow sufficient reactivity to include any arbovirosis on the territories of Mayotte and La Réunion.

ELIGIBILITY:
1st case :

Inclusion Criteria:

* Adult, child or newborn > 2.5kg on day of inclusion.
* Use of one of the hospital departments participating in the research, in an emergency room, full hospitalization, day hospitalization or outpatient clinic.
* Suspected, probable or biologically confirmed arbovirosis:

A suspected case of arbovirosis is defined as :

* asymptomatic contact case of a patient with probable or confirmed arbovirosis
* symptomatic or non-symptomatic newborns of mothers who were viremic for arbovirosis during pregnancy, or who had probable or confirmed arbovirosis during pregnancy.
* In a patient with a history of a stay in an arbovirus circulation zone in the 2 weeks prior to consultation (for imported cases only).
* In a patient with compatible clinical symptoms during the epidemic period

A probable case of arbovirosis is defined by :

* the association of at least 2 objectified or reported signs or biology suggestive of arbovirosis: fever (reported by the patient or family, or documented), headache, rash, myalgias, arthralgias, abdominal pain, bleeding, thrombocytopenia, or
* for children under 6: by the reporting (by the family or documented) of a fever on the day of inclusion or in the preceding 7 days, possibly accompanied by pain.

A biologically confirmed case of arbovirosis is defined by :

- A positive plasma RT-PCR or urine RT-PCR (Zika virus)

Case 2 : - Retrospectively, patients with sufficiently documented definite, probable or suspected arbovirosis, who give oral consent for their data to be collected retrospectively and/or to continue the study follow-up.

Exclusion Criteria:

1. Patient ou titulaire de l'autorité parentale non affiliés ou non bénéficiaires d'un régime de sécurité sociale.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2037-05-05 (Estimated); Study Completion 2037-05-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a severe form of arbovirosis | THROUGHT STUDY COMPLETION AN AVERAGE OF 3 YEARS
  Occurrence of a severe form of arbovirosis: shock, internal hemorrhage, severe organ failure (visceral, cardiac, neurological, ophthalmological, renal, pulmonary, hepatic, etc.), death caused directly or indirectly by the infection.

CONTACTS AND LOCATIONS:
Locations (1):
- PRCT, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No